CLINICAL TRIAL: NCT04820296
Title: Effects of Solution-Oriented Approach Applied to Primigravidas on Psychosocial Health, Fear of Childbirth and Postnatal Senses of Security: A Randomized Controlled Study
Brief Title: Effects of Solution-Oriented Approach on Psychosocial Health, Fear of Childbirth and Postnatal Senses of Security
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yeşim Anık, Research Assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Necmettin EU
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Fear of Childbirth; Psychosocial Health; Pregnancy; Postpartum; Childbirth
Keywords: Solution-oriented approach; Fear of childbirth; Psychosocial health; mothers; Feelings of security; Pregnancy

STUDY DESIGN:
Intervention Model Description: Posttest and control grouped randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Pregnant women in the experimental group will be given 4 sessions Solution-Oriented Approach program, starting at the 32th week of pregnancy. Pregnants in the experimental group will be administered the Wijma Birth Expectation/Experience Scale (W-DEQ-A) and Pregnancy Psychosocial Health Assessment Scale (PPHAS) before the intervention. After the program is completed, a training booklet will be provided for pregnant women and (W-DEQ-A) and PPHAS will be applied again. With pregnant women, 37-40. between gestational weeks, they will be contacted again, face-to-face interview method (W-DEQ-A) and PPHAS again will be evaluated. The pregnant women will inform the researcher by phone after the delivery and the researcher will visit the hospital within the first 24 hours after the delivery to evaluate the mothers' birth fear levels Scale (W-DEQ-B). At the end of the first postpartum week, the postnatal senses of security of the mothers will be evaluated by telephone follow-up counseling.
  Interventions: Other: Solution-Oriented Approach
- Control group (No Intervention): Pregnant women in the control group will only receive routine care. Pregnant women in the control group will be administered the same scales simultaneously with the experimental group.

INTERVENTIONS:
Other: Solution-Oriented Approach — First Session: Sharing thoughts about perception of childbirth, Creating positive goals, Informing about Birth, Birth Process, Basic Breathing Exercises and Deep Relaxation Exercises, Homework Second Session: Evaluating homework, Sharing thoughts about fear of childbirth, Miracle Question Technique, Evaluating with the Rating Questions Technique, Reframing the problem, Briefing on 'Body-Mind Connection at Birth, Fear-Tension-Pain Cycle, Hormones of Birth' and Breathing exercises, Homework Third session: Evaluating homework, Sharing thoughts about positive birth story, Information on symptoms indicating that the childbirth is approaching, pushing techniques, delivery positions, endorphin massage and breathing exercises (4/8 breaths, full breath when baby moves), Homework Fourth Session: Evaluating homework, Mother Baby Friendly Caesarean and Breathing exercises (3 candles a feather breath), Sharing feelings about the counseling process
  Arms: Experimental group

SUMMARY:
This study was planned as a randomized controlled experimental study with posttest and control group in order to evaluate the effect of the solution focused approach method applied to primigravidas on psychosocial health, fear of childbirth and postnatal security sensations

DETAILED DESCRIPTION:
Pregnancy and childbirth process is a natural life event for women, as well as a period of physiological, psychological and social changes. Biopsychosocial changes experienced during this period increase the risk of encountering factors that may cause anxiety and stress. For this reason, psychosocial health can be negatively affected during pregnancy. One of the most important factors threatening psychosocial health during pregnancy is the fear of childbirth. Fear of childbirth emerges especially in the last trimester, causing the woman to spend the unique and special pregnancy process in restlessness and tension. Fear of childbirth may cause consequences such as preferring not to pregnant, as well as bring about complications related to the childbirth process and postpartum period. Within the scope of studies to manage the fear of childbirth, many approaches are used, such as childbirth preparation classes, breathing techniques, hydrotherapy, hypnosis, doula support, holistic care and support, cognitive and behavioral therapies, psychoeducation. One of the most current methods used in the management of childbirth fear is solution-oriented approach. Solution Focused Approach leads the individual to solution again and again instead of focusing on solving the problem as a separate method, it offers an approach focused on the solution itself. It is stated that the philosophy of solution-oriented approach in line with the individual-centered perspective, principles and values is compatible with the basic value and philosophy of nursing. As a result of the studies, it has been determined that the solution-oriented approach method is a shorter-term and effective counseling approach compared to other alternative approaches, after the approach, improvement / decrease in related behavioral problems is observed and it provides significant positive benefits. It is also stated to be more economical due to its wide application areas. This study was planned as a randomized controlled experimental study with posttest and control group in order to evaluate the effect of the solution focused approach method applied to primigravidas on psychosocial health, fear of childbirth and postnatal security sensations.

Preliminary evaluation in the study will be made in the pregnant policlinic of a university hospital in the city center of Konya. Verbal and written permission will be obtained from pregnant women who meet the inclusion criteria according to the result of the preliminary evaluation made in the outpatient clinic. For the sample calculation of the study, an experimental study evaluating the effect of childbirth preparation education on the fear of childbirth, postpartum self-efficacy and posttraumatic stress disorder was taken as reference. The sample calculation of the research was made in G * Power (3.1.9.2) program. In the calculation based on the reference study data (90% power, effect size 0.96, alpha level 0.05, beta level 0.90), it was found that a total of 48 cases, 24 for the experimental group and 24 for the control group, were suitable for statistical analysis.

In the literature, it has been determined in the experimental studies on this issue that there is loss of subjects between 10% and 40%. In this study, considering the loss rates in the literature, assuming that there would be 40% loss, it was decided to take 68 pregnant women, 34 to the experimental group and 34 to the control group. Pregnant women included in the research will be assigned to the experimental and control groups by block randomization method according to the randomization list.

In the collection of the data,

* The introductory information form developed by the researcher using the literature,
* The Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ version A and B)
* Psychosocial Health Assessment Scale in Pregnancy,
* The Mother's Postnatal Sense of Security Scale will be used.

İmplementation of the Research

Four sessions (one session per week) Solution Focused Approach program will be applied to the pregnants in the experimental group. The duration of each session is planned as 60 minutes. The program will be implemented in groups of five. The first session will start at the 32nd week of pregnancy, and the program will be completed at the end of the 35th week of pregnancy. After the program is completed, a training booklet prepared by the researcher will be given to the pregnant women in the experimental group so that they can repeat the information they have learned until delivery. After the training program is completed (WDEQ) version A and Psychosocial Health Assessment Scale in Pregnancy will be applied again (2nd measurement).With pregnant women, 37-40. between gestational weeks, they will be contacted again, and when they come to the hospital for routine pregnancy follow-up, face-to-face interview method (WDEQ) version A and Psychosocial Health Assessment Scale in Pregnancy (3rd measurement) again will be evaluated. The pregnant women will inform the researcher by phone after the delivery and the researcher will visit the hospital within the first 24 hours after the delivery to evaluate the mothers' birth fear levels (WDEQ) version B (only the posttest). At the end of the first postpartum week, the postnatal senses of security of the mothers (only post-test) will be evaluated by telephone follow-up counseling.

Evaluation of the Data

Coding and evaluation of data will be done in computer environment with SPSS 22.0 (Statistical Program for Social Sciences) package program. The suitability of the research data to normal distribution will be determined by Kolmogorov-Smirnov test with Lilliefor, normal distribution curve, Skewness and Kurtosis test. Descriptive statistics will be evaluated by the number, percentage, average and standard deviation. For the implementation of the study, the ethics committee permission numbered 2020/2352 was obtained from Necmettin Erbakan University Meram Medical Faculty Pharmaceuticals and Non-Medical Research Ethics Committee and the institutional permission numbered E.33709 from Necmettin Erbakan University Meram Medical Faculty Hospital Chief Physician. Pregnant women who will be included in the research sample will be informed before the study that the purpose of the study and participation in the study is in line with the principle of volunteering, and "Informing and Consent of Volunteers Consent Form" will be signed.

Dependent Variables

* Pregnant women (W-DEQ) A version scale mean scores,
* Pregnant women (W-DEQ) B version scale mean scores,
* Psychosocial Health Assessment Scale in Pregnancy mean scores,
* The mean scores of the Postnatal Sense of Security Scale of the pregnant women.

Independent variable

• Solution Focused Approach Program

ELIGIBILITY:
Inclusion Criteria:

* At least primary education graduate
* Speaking and understanding Turkish
* Pregnant women between the ages of 18-35
* Residing at the provincial border of Konya
* Primigravidas
* Women who got pregnant without treatment pregnancy,
* Have no barriers to vaginal birth,
* Pregnant women who are at the 32nd gestational week according to their last menstrual week
* Pregnant women with a single and healthy fetus

Exclusion Criteria:

* Pregnant women with any risky pregnancy history (Placenta previa, preeclampsia, oligohydramnios and polyhydramnios, gestational diabetes etc.),
* Pregnant women with any systemic and neurological disease,
* Pregnant women with chronic and/or psychiatric health problems (based on self-report and clinical diagnosis),
* Pregnant women with cesarean indication,
* Pregnant women participating in any birth preparation training program.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Enrollment: 68 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Wijma Birth Expectancy / Experience Scale (W-DEQ) Version A | First assessment will be made at the baseline (pre-intervention).
  It is a Likert-type scale consisting of 33 items and 6 sub-dimensions that measure stress and fear during birth. The validity and reliability study of the scale was conducted by Körükcü et al. (2012). The first sub-dimension will determine the thoughts about childbirth contractions and how the birth will be in general, the second sub-dimension will determine the characteristics of childbirth contractions and the characteristics of contractions felt during childbirth, the third sub-dimension will determine what the woman will feel during childbirth, the fourth sub-dimension will determine what the woman will be when the contractions are most intense. The fifth sub-dimension consists of questions about the emotions imagined at the birth of the baby, and the sixth dimension consists of questions for evaluating the woman's thoughts about childbirth and delivery in the last month. Answers in the scale are scored between 0 and 5. Higher item total score indicates high level of fear.
Wijma Birth Expectancy / Experience Scale (W-DEQ) Version A | The second assessment will take place 4 weeks after the first assessment (after the program is completed).
  It is a Likert-type scale consisting of 33 items and 6 sub-dimensions that measure stress and fear during birth. The validity and reliability study of the scale was conducted by Körükcü et al. (2012). The first sub-dimension will determine the thoughts about childbirth contractions and how the birth will be in general, the second sub-dimension will determine the characteristics of childbirth contractions and the characteristics of contractions felt during childbirth, the third sub-dimension will determine what the woman will feel during childbirth, the fourth sub-dimension will determine what the woman will be when the contractions are most intense. The fifth sub-dimension consists of questions about the emotions imagined at the birth of the baby, and the sixth dimension consists of questions for evaluating the woman's thoughts about childbirth and delivery in the last month. Answers in the scale are scored between 0 and 5. Higher item total score indicates high level of fear.
Wijma Birth Expectancy / Experience Scale (W-DEQ) Version A | Third assessment will take place average 3 weeks after the second assessment.
  It is a Likert-type scale consisting of 33 items and 6 sub-dimensions that measure stress and fear during birth. The validity and reliability study of the scale was conducted by Körükcü et al. (2012). The first sub-dimension will determine the thoughts about childbirth contractions and how the birth will be in general, the second sub-dimension will determine the characteristics of childbirth contractions and the characteristics of contractions felt during childbirth, the third sub-dimension will determine what the woman will feel during childbirth, the fourth sub-dimension will determine what the woman will be when the contractions are most intense. The fifth sub-dimension consists of questions about the emotions imagined at the birth of the baby, and the sixth dimension consists of questions for evaluating the woman's thoughts about childbirth and delivery in the last month. Answers in the scale are scored between 0 and 5. Higher item total score indicates high level of fear.
Wijma Birth Expectancy / Experience Scale (W-DEQ) Version B | The W-DEQ scale version B (only posttest) will be administered within the first 24 hours of postpartum.
  W-DEQ version B was developed by Klaas and Barbro Wijma (1998) to measure the experiences of women with fear of childbirth in the postpartum period. Körükcü et al. (2014), the scale, which was adapted to Turkish and valid and reliable, consists of 32 items and six sub-dimensions. The sub-dimensions of the scale are, respectively, anxiety about labor pain, inadequacy of positive behavior, loneliness, inadequate positive emotions, anxiety about delivery, and anxiety about the baby. Answers in the scale are scored between 0 and 5. While the minimum score in the scale is 0, the maximum score is 160. As the score increases, the fear of childbirth that women experience increases.

SECONDARY OUTCOMES:
Psychosocial Health Assessment Scale During Pregnancy | First assessment will be made at the baseline (pre-intervention).
  The scale, which was developed by Yıldız (2011) and whose validity and reliability was made, evaluates psychosocial health during pregnancy as a whole. It is a 5-point Likert-type scale consisting of a total of 46 items and 6 sub-dimensions. The sub-dimensions of the scale include the Features of Pregnancy and Spousal Relationship, Features of Anxiety and Stress, Characteristics of Domestic Violence, Features of Psychosocial Support Requirement, Family Features and Physical-Psychosocial Changes Related to Pregnancy. In this scale, the lowest score that can be taken in total is 46, the highest score is 230. The average value is determined by dividing the total score determined in the scale by the number of items and is scored between 1 and 5. "1" indicates that psychosocial health is very bad and "5" indicates that it is very good, and the evaluation is interpreted in that context whichever direction the scores approach.
Psychosocial Health Assessment Scale During Pregnancy | The second assessment will take place 4 weeks after the first assessment (after the program is completed).
  The scale, which was developed by Yıldız (2011) and whose validity and reliability was made, evaluates psychosocial health during pregnancy as a whole. It is a 5-point Likert-type scale consisting of a total of 46 items and 6 sub-dimensions. The sub-dimensions of the scale include the Features of Pregnancy and Spousal Relationship, Features of Anxiety and Stress, Characteristics of Domestic Violence, Features of Psychosocial Support Requirement, Family Features and Physical-Psychosocial Changes Related to Pregnancy. In this scale, the lowest score that can be taken in total is 46, the highest score is 230. The average value is determined by dividing the total score determined in the scale by the number of items and is scored between 1 and 5. "1" indicates that psychosocial health is very bad and "5" indicates that it is very good, and the evaluation is interpreted in that context whichever direction the scores approach.
Psychosocial Health Assessment Scale During Pregnancy | Third assessment will take place average 3 weeks after the second assessment.
  The scale, which was developed by Yıldız (2011) and whose validity and reliability was made, evaluates psychosocial health during pregnancy as a whole. It is a 5-point Likert-type scale consisting of a total of 46 items and 6 sub-dimensions. The sub-dimensions of the scale include the Features of Pregnancy and Spousal Relationship, Features of Anxiety and Stress, Characteristics of Domestic Violence, Features of Psychosocial Support Requirement, Family Features and Physical-Psychosocial Changes Related to Pregnancy. In this scale, the lowest score that can be taken in total is 46, the highest score is 230. The average value is determined by dividing the total score determined in the scale by the number of items and is scored between 1 and 5. "1" indicates that psychosocial health is very bad and "5" indicates that it is very good, and the evaluation is interpreted in that context whichever direction the scores approach.
Mother's Postnatal Senses of Security Scale | At the end of the 7th postpartum day, follow-up counseling will be provided by telephone and the Postpartum Sense of Security Scale (posttest only) will be filled.
  Postpartum Security Feelings Scale was developed by Eva K Persson et al. (2007) to determine mothers' sense of security in the first week after birth. Scale Geçkil et al. Its validity and reliability study was carried out by adapting it to Turkish in 2016. The scale is in the form of a 4-point Likert consisting of 18 items and 4 sub-dimensions. The lowest score that the participants can get from the total of the scale is 18 and the highest score is 72. 4 sub-dimensions of the scale; "Reinforcing Behavior" consists of "General Goodness", "Family Ties" and "Breastfeeding Behavior" dimensions. High scores indicate that mothers have a good sense of security in their postpartum period (Geçkil et al.2016).

CONTACTS AND LOCATIONS:
Overall Officials: YEŞİM ANIK, MSc, Principal Investigator — Necmettin Erbakan University; KAMİLE ALTUNTUĞ, PhD, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: The study protocol will be published in a peer-reviewed journal within 6 months.
Access Criteria: After the study protocol is published, the name and link of the journal in which the publication was published will be shared.